# The Add-On Effect of Lactobacillus plantarum PS128 in Patients With Parkinson's Disease: A Pilot Study

## NCT04389762

# **December 31, 2021**

#### 1. Assessment of Outcomes

In this study, the primary measurements were the Unified Parkinson's Disease Rating Scale part III (UPDRS-III) motor scores and changes in patient's "ON-OFF" diary recordings, and modified Hoehn and Yahr scale (mHYS). The secondary measurements were the 39-item Parkinson's Disease Questionnaire (PDQ-39), Non-Motor Symptoms Scale (NMSS), BDI-II, patient assessment of constipation symptoms (PAC-SYM), Patient Global Impression of Change (PGI-C), and other metabolic profiles. All clinical assessments were performed after 12 h of overnight withdrawal from antiparkinsonian medications (24 h of withdrawal was needed if the participants were taking prolonged release dopaminergic agonists). Therefore, UPDRS-III and mHYS were scored in the OFF state the next morning as well as the metabolic profiles. Then, the medications were self-administered by each patient before the secondary measurements. The UPDRS, mHYS, PDQ-39, NMSS, BDI-II, PAC-SYM, and PGI-C were scored 40-60min later in the patients' best ON state. For safety assessment, physical and neurological examinations were performed to evaluate the overall health of the subjects at weeks 0 and 12. In addition, all subjects were actively monitored for the occurrence of adverse events by telephone at least once per week.

### 2. Biochemical Measurements

A blood sample of 15mL and a urine sample of 10mL were collected at weeks 0 and 12. The serum high-sensitivity C-reactive protein level was determined by turbidimetric immunoassay. The plasma myeloperoxidase (MPO) and urinary 8-hydroxy-2'-deoxyguanosine were measured by enzyme-linked immunosorbent assay. The plasma glutathione peroxidase and total antioxidant capacity were measured by Ransel test kits (Randox Laboratories Ltd., UK) and ferric-reducing ability, respectively. The urinary creatinine (CRE) level was determined by MeDiPro creatinine test. All procedures were performed according to the manufacturer's

instructions.

# 3. Statistics Analysis

For this clinical trial, all statistical analyses are conducted using SPSS software (Version 22.0, IBM Corp., Armonk, NY). Descriptive statistics are presented as mean  $\pm$  standard deviation (SD). The Wilcoxon signed-rank test is used for comparisons on ordinal scales when a significant difference is observed. This test is employed to evaluate changes in total UPDRS, UPDRS-I, UPDRS-II, UPDRS-III, UPDRS-IV, as well as subscores for tremor, rigidity, akinesia, and postural instability gait disorder (PIGD), mHYS, diary recordings, PDQ-39, BDI-II, and PAC-SYM from baseline (V0) to post-intervention (V1, 12 weeks). Effect sizes are calculated using Cohen's d, defined as the mean change divided by the SD. For nominal scale variables with significant differences, the chi-square test is applied, particularly for the NMSS. Paired Student's t-test is used to assess differences in metabolic parameters between baseline and after the probiotics intervention. All data are reported as the mean  $\pm$  SD, with statistical significance set at p < 0.05.